CLINICAL TRIAL: NCT07137845
Title: Virtual Reality and Cranial Nerve Non-invasive Neuromodulation to Improve Quality of Life for Veterans Living With Post-traumatic Stress Disorder and Chronic Pain
Brief Title: Virtual Reality and Cranial Nerve Non-invasive Neuromodulation to Improve Quality of Life for Veterans
Acronym: VR & CN-NINM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Chronic Pain Center of Excellence for Canadian Veterans (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2026-5892
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; PTSD - Post Traumatic Stress Disorder; Quality of Life (QOL)
Keywords: Chronic pain; PTSD; Veterans; Autonomic nervous system; Virtual reality (VR); Cranial nerve non-invasive neuromodulation (CN-NINM); Quality of life
MeSH Terms: conditions — Chronic Pain; Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study model is a randomized controlled feasibility study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (VR) + Cranial nerve non-invasive neuromodulation (CN-NINM) (Experimental): CN-NINM will be applied during the VR interventions (20 min).
  Interventions: Procedure: Virtual reality; Procedure: Cranial nerve non-invasive neuromodulation (CN-NINM)
- Virtual reality (VR) + sham CN-NINM (Experimental): Sham CN-NINM (no stimulation) will be applied during the VR interventions (20 min).
  Interventions: Procedure: Virtual reality; Procedure: Sham CN-NINM

INTERVENTIONS:
Procedure: Virtual reality — The VR intervention will take place in a quiet room. The participant will be installed in a seated position, wearing a virtual reality headset that includes an audio device playing sounds. The eyes are covered by a mask featuring a screen showing calming 3D VR images (e.g. beach landscapes), designed by our team. The intervention lasts 20 minutes. The hypnotic suggestions with auditory and visual calming stimulations will help the person to focus on the present moment, to reduce anxiety and painful sensations.
Procedure: Cranial nerve non-invasive neuromodulation (CN-NINM) — During each intervention including CN-NINM, this latter will be applied for 20 minutes, with the help of a portable stimulator comprising a network of 18 electrodes, directly on the tongue of the participants. The participants will hold the CN-NINM in place by pressing their tongue upwards. The CN-NINM will generate high-frequency pulses (50 µsec to 150 Hz), and the intensity of the stimulus will be set by each participant to a comfortable level of sensation, similar to the sensation in the mouth of a soft drink.
  Arms: Virtual reality (VR) + Cranial nerve non-invasive neuromodulation (CN-NINM)
Procedure: Sham CN-NINM — In this study, we will have a control intervention which will be placebo CN-NINM. For placebo CN-NINM, participants will wear the device such as the real CN-NINM group, without having experienced the tingling sensation beforehand, so they will not know what the CN-NINM potential effect is.
  Arms: Virtual reality (VR) + sham CN-NINM

SUMMARY:
Veterans in Canada are twice as likely as the general population to experience chronic pain. This pain is often linked to post-traumatic stress disorder (PTSD), and both have a major impact on their quality of life. The autonomic nervous system (ANS) plays a key role in these pathologies, making its modulation a promising therapeutic target. Veterans are already experiencing pain and PTSD relief via virtual reality (VR), mostly through ANS reactivity modulation. Long-term exposure (desensitization) and the calming effect are the two forms of VR; the latter is more tolerable and more suited for ANS rebalance. Its benefits on pain, however, are still mild and transient. In order to further enhance these benefits, cranial nerve non-invasive neuromodulation (CN-NINM), a novel technology that enables the direct flow of neuronal impulses through tongue stimulation, is suggested to be combined with virtual reality (VR). The goal of this project is to document the feasibility of an intervention combining virtual reality (VR) with real and sham cranial nerve non-invasive neuromodulation (CN-NINM) in veterans with post-traumatic stress disorder and chronic pain.

The secondary objectives are: 1) to explore and compare the effect of the two interventions (VR + real CN-NINM vs. VR + sham CN-NINM) on various clinical measures, and 2) to explore and compare the effect of these two interventions on autonomic nervous system (ANS) activity.

Each intervention will be applied for 20 minutes. Their painful condition (whether diagnosed or not, type, location, intensity, and unpleasant aspects of the pain) as well as their PTSD-related symptoms will be assessed before and after the intervention.

At the end of this study, it is expected that the CN-NINM could become a complementary treatment option for relieving pain and PTSD symptoms in PVs and, ultimately, improving their quality of life.

DETAILED DESCRIPTION:
In Canada, many veterans suffer from chronic pain, with a prevalence twice that of the general population. Chronic pain is often linked to post-traumatic stress disorder (PTSD), and both conditions impact the functioning and quality of life of veterans. Recent studies suggest that the autonomic nervous system (ANS) plays an important role in the pathophysiology of chronic pain and PTSD, making it a therapeutic target of choice.

Virtual reality (VR) is an approach already used with this population, and its effectiveness in relieving pain and PTSD is well documented in veterans, mainly through modulation of ANS activity. Two VR approaches are commonly used: prolonged exposure VR (desensitization) and calming VR (aimed at normalizing the stress response and ANS activity). Calming VR is better tolerated than prolonged exposure VR and remains better suited to rebalancing ANS activity and relieving symptoms. It helps calm the ANS and relieve pain (acute and chronic) when combined with traditional rehabilitation, but its effects on pain intensity remain modest and limited in time.

To enhance the benefits of VR, the investigators suggest combining VR with a non-pharmacological approach, as recommended by experts. This approach is known as non-invasive cranial nerve neuromodulation (CN-NINM). CN-NINM is an innovative approach that stimulates the cranial nerves via electrodes placed directly on the tongue; the impulses reach and modulate the activity of the ANS structures located in the brainstem. These structures are linked to autonomic functions and pain modulation. This combination could reinforce and prolong the positive effects of VR on pain in veterans.

Primary objective: To document the feasibility of an intervention combining virtual reality (VR) with real and sham non-invasive cranial nerve neuromodulation (CN-NINM) in veterans with post-traumatic stress disorder and chronic pain.

Secondary objectives : 1) to explore and compare the effect of the two interventions (VR + real CN-NINM vs. VR + sham CN-NINM) on the following clinical measures: i) quality of life, ii) pain (e.g., intensity, impact on physical function), and iii) PTSD-related symptoms, 2) to explore and compare the effect of these two interventions on autonomic nervous system (ANS) activity, and 3) to determine whether there are associations between changes in quality of life and clinical changes on the one hand, and physiological changes (autonomic nervous system activity) on the other.

Methods: To do this, the investigators propose a feasibility study with two groups (experimental group vs. control group) with 30 participants. Participants will take part in an assessment of their pain condition (diagnosed or undiagnosed pain condition, type, location, intensity, and unpleasant aspects of pain) and their PTSD-related symptoms. The participants will also complete clinical questionnaires assessing their pain, PTSD-related symptoms, and their impact on physical function and quality of life. The investigators will also take various autonomic measurements (blood pressure, heart rate variability [HRV], electrodermal response) to characterize autonomic nervous system activity. Sociodemographic, pain and PTSD-related variables will be collected to confirm participant eligibility.

Participants will come to the laboratory eight times to receive the interventions (VR + real CN-NINM or VR + sham CN-NINM) and will complete online questionnaires at four measurement points (T0, T1, T2, and T3). Participants will be seated and wearing a virtual reality headset equipped with an audio device that plays sounds. The VR headset will broadcast calming images designed by our team specifically for veterans for 20 minutes. CN-NINM will be applied using a portable stimulator directly to participants' tongues for 20 minutes, at the same time as the VR. For the control group, participants will apply CN-NINM to their tongues without any perceptible stimulus.

ELIGIBILITY:
Inclusion Criteria:

1. Be a veteran;
2. Be ≥18 years old;
3. Have a diagnosis of chronic musculoskeletal pain (pain > 6 months);
4. Have been diagnosed with PTSD by a health professional and/or have a PTSD Checklist for DSM-5 (PCL-5) score > 30/80 and
5. Speak English or French.

Exclusion Criteria:

1. Bipolar disorder, psychosis;
2. Neuropathic pain (based on the Neuropathic Pain Diagnosis and Questionnaire (DN4));
3. Visual disorders or photosensitivity, color blindness;
4. Epilepsy, motion sickness and
5. Any containdications to CN-NINM.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate for the project | Information will be assessed at the end of the recruitment period, at week 28.
  This outcome will be compiled by the total number of participants recruited, divided by the average number of months recruiting.
Refusal to participate and the reasons | Information will be assessed throughout the project recruitment period (average of 7 months).
  Participant refusal will be quantified by recording the number of individuals who declined to take part in the study. The reasons for refusal will also be documented.
Dropped out rate of the project in percent | Information will be assessed through project completion, an average of 9 months.
  The dropout rate will be determined by calculating the proportion of participants who discontinued their participation relative to the total number of participants initially enrolled, expressed as a percentage.
Adherence to the interventions (VR + CN-NINM, VR + CN-NINM sham) in percent | Information will be assessed through study completion, an average of 9 months.
  Adherence to interventions will be calculated by the number of visits completed out of the total number expected X 100%, by attrition and loss to follow-up.
Safety-related informations for each intervention as assessed by a questionnaire | Information will be assessed through study completion, an average of 9 months.
  Safety-related informations for each intervention will be assessed with a questionnaire that will provide a number and percentage of participants who have experienced adverse events (frequency, type and severity of adverse events).

SECONDARY OUTCOMES:
Change in measures of blood pressure | The assessments will be done at baseline and just after the 20 minutes application of each intervention (VR + CN-NINM, VR+CN-NINM sham).
  Change in measures of blood pressure will be assessed with NIBP100E Finger Cuff Sensors and Blood Pressure Cuff from BIOPAC.
Change in heart rate variability | The assessments will be done at the baseline, during the 20 minutes of application of each intervention (VR + CN-NINM, VR+CN-NINM placebo) and just after the 20 minutes of applications of each intervention (VR + CN-NINM, VR+CN-NINM placebo).
  Change in heart rate variability will be assessed with ECG Electrocardiogram Amplifier (MP200) from BIOPAC. Investigators will look at: - Root Mean Square of Successive Differences or RMSSD (measurement that reflects the activity of the parasympathetic nervous system), - High Frequencies or HF (representing the activity of the parasympathetic nervous system) and - Low Frequencies/High Frequencies [LF/HF] ratio (indicator of the balance between the activity of the sympathetic nervous system (SNS) and the parasympathetic nervous system (SNP)).
Change in electrodermal activity response | The assessments will be done at the baseline, during the 20 minutes application of each intervention (VR + CN-NINM, VR+CN-NINM placebo) and just after the 20 minutes application of each intervention (VR + CN-NINM, VR+CN-NINM placebo).
  Change in electrodermal activity (microsiemens) will be assessed with the EDA finger transducer from BIOPAC.
Change in pain intensity and impact on physical function using the Brief Pain Inventory (BPI) | The questionnaire will be done at the baseline (T0), just after the 8 weeks of each intervention (VR + CN-NINM, VR+CN-NINM placebo) (T1), one month (T2) and three month (T3) after the last intervention.
  Change in pain intensity and impact will be assessed using a scored questionnaire. The questionnaire score is divided into two dimensions: the pain impact on physical function score (/70) and the severity score (/40). A high score would indicate severe pain with a significant impact on physical function.
Change in the qualitative aspect of pain with the McGill Pain Questionnaire (MPQ) | The questionnaire will be done at the baseline (T0), just after the 8 weeks of each intervention (VR + CN-NINM, VR+CN-NINM placebo) (T1), one month (T2) and three month (T3) after the last intervention.
  Change in the qualitative aspect of pain will be measured with the McGill Pain Questionnaire, a scored multi-dimensional questionnaire. The questionnaire score range from 0 (no pain) to 78 (severe pain). A higher total score indicates a more intense pain experience.
Change in pain-related disability using the Pain Disability Questionnaire (PDQ) | The questionnaire will be done at the baseline (T0), just after the 8 weeks of each intervention (VR + CN-NINM, VR+CN-NINM placebo) (T1), one month (T2) and three month (T3) after the last intervention.
  Change in pain-related disability will be evaluated using the PDQ. The total PDQ score range from 0 to 150. A high score indicates more pain-related disability.
Change in Patient Global Impression of Change (PGIC) | The questionnaire will be done at the baseline (T0), just after the 8 weeks of each intervention (VR + CN-NINM, VR+CN-NINM placebo) (T1), one month (T2) and three month (T3) after the last intervention.
  The PGIC is a self-report scale used to measure a person's impression of the effectiveness of a treatment or intervention. It is a 7-point scale on which patients rate their overall change, with scores ranging from "very much improved," to "very much worse".
Change in Post-traumatic Stress Disorder Checklist - V (PCL-V) | The questionnaire will be done at the baseline (T0), just after the 8 weeks of each intervention (VR + CN-NINM, VR+CN-NINM placebo) (T1), one month (T2) and three month (T3) after the last intervention.
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including: monitoring symptom change during and after treatment, screening individuals for PTSD and making a provisional PTSD diagnosis. A total symptom severity score (ranging from 0 to 80) can be obtained by summing the scores for each of the 20 items.
Change in Composite Autonomic Symptom Scores - 31 (COMPASS-31) | The questionnaire will be done at the baseline (T0), just after the 8 weeks of each intervention (VR + CN-NINM, VR+CN-NINM placebo) (T1), one month (T2) and three month (T3) after the last intervention.
  The COMPASS-31 is a self-report questionnaire used to evaluate the severity of autnomic nervous system (ANS) dysfunction. It consists of 31 items across six domains and provides a weighted total score (ranging from 0 to 100), with higher scores indicating greater autonomic dysfunction.
Change in the quality of life with Veterans 36-item Short Form Survey (Veterans SF-36) | The questionnaire will be done at the baseline (T0), just after the 8 weeks of each intervention (VR + CN-NINM, VR+CN-NINM placebo) (T1), one month (T2) and three month (T3) after the last intervention.
  The Veterans SF-36 is a self-administered health assessment tool used to evaluate the health-related quality of life of veterans. The Veterans SF-36 measures eight dimensions of health status including physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, energy/fatigue, social functioning, role limitations due to emotional problems, and mental health. Each domain's raw scores are standardized to a 0-100 scale for scoring, where higher scores denote greater health.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Léonard, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement (CdRV), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No